CLINICAL TRIAL: NCT06310915
Title: This Study is a Pilot Study in Driver-negative Locally Advanced/Late-stage Nonsmall Cell Lung Cancer With ECOG PS=2 Analysing the Efficacy, Safety and Efficacy of Oral Chemotherapy in Combination With PD-1 Inhibitors and Safety of Oral Chemotherapy in Combination With PD-1 Inhibitors in Patients With Locally Advanced/Advanced Non-cellular Lung Cancer withECOG PS=2.This is a Prospective, Single-arm, Multicentre, Observational Study
Brief Title: Oral Chemotherapeutic Drugs Were Analyzed in Patients With Driver Gene Negative Locally Advanced/Advanced Non-small Cell Lung Cancer With PS Score 2 A Prospective, Single-arm, Multicenter, Observational Study on the Efficacy and Safety of Radiochemotherapy Combined With PD-1 Inhibitor
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Guangzhou Institute of Respiratory Disease
Other Study IDs: CROC202310
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB/IV
Keywords: Advanced non-small cell lung cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Navelbine oral,Pembrolizumab — Oral vinorelbine was administered three times weekly, and pembrolizumab was administered every 3 weeks

SUMMARY:
Oral chemotherapeutic drugs were analyzed in patients with driver gene negative locally advanced/advanced non-small cell lung cancer with PS score 2 A prospective, single-arm, multicenter, observational study on the efficacy and safety of radiochemotherapy combined with PD-1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of 18-80 years old, both sexes;
* 2. Patients with histologically confirmed advanced non-small cell lung cancer with stage IIIB /IV disease (according to the International Association for the Study of Lung Cancer Staging Manual for Thoracic Tumors, 8th edition) or disease recurrence or progression after multimodal treatment (radiotherapy, surgical resection, or definitive chemoradiotherapy for locally advanced disease);
* 3. Patients should have no EGFR gene sensitive mutations (including but not limited to exon 19 deletion, exon 21 L858R mutation, exon 21 L861Q, exon 18 G719X, or exon 20 S768I mutation), ALK gene rearrangement, or ROS1;

Exclusion Criteria:

* 4.Participants had to have measurable lesions on CT or MRI according to RECIST 1.1 (tumor imaging was performed within 28 days before the first dose of study drug) or clinically significant lesions that could be followed for response according to RECIST 1.1 by the investigator;
* 5. No prior systemic therapy (patients with prior platinum-based adjuvant chemotherapy, neoadjuvant chemotherapy, or definitive chemoradiotherapy for advanced disease could enter if disease progression occurred >6 months after the last treatment);
* 6. Ecog ps =2分;
* 7. Estimated survival time > 12 weeks;

exclusion criteria:

* 1. Subjects requiring systemic treatment with glucocorticoids (>10mg prednisone equivalent daily) or other immunosuppressive drugs within 14 days before the first dose of study drug were excluded. Subjects using inhaled or topical corticosteroids, as well as adrenocortical steroid replacement therapy doses equivalent to >10 mg prednisone/day, were eligible to participate if they did not have active autoimmune disease. In addition, the participants had to have discontinued glucocorticoids or were taking prednisone at a dose of less than 10mg per day (or equivalent) that was stable or reduced.
* 2. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies or any other antibody or agent that targets T-cell costimulation or the immune checkpoint pathway;
* 3. Previous treatment with a trial drug;
* 4. Subjects with active CNS metastases were excluded. Participants could participate if CNS metastases could be adequately treated and if their neurologic symptoms (other than residual signs or symptoms related to CNS therapy) returned to baseline at least 2 weeks before enrollment.
* 5. Previous malignant tumor (excluding non-melanoma skin cancer and the following carcinomas in situ: Cancer in situ of the bladder, stomach, colon, endometrium, cervix/dysplasia, melanoma, or breast) were excluded unless they had achieved a complete response at least 2 years before study entry and had not undertaken and did not require additional therapy (other than antiestrogen/androgen therapy or bisphosphonate therapy) during the study. Subjects with other active malignant tumors requiring concurrent treatment were excluded.
* 6. Women with a positive pregnancy test at recruitment or before study dosing;
* 7. Carcinomatous meningitis;
* 8. The subject has a history of interstitial lung disease (e.g., sarcoidosis) that is symptomatic or may preclude the detection or management of suspected drug-related pulmonary toxicity;
* 9. Subjects with COPD can be enrolled in the study if the disease is controlled at the time of enrollment;
* 10. Serious or uncontrolled illness that, in the opinion of the investigator, would increase the risk associated with participation in the study or administration of the study drug, affect the ability of the subject to receive the treatment specified in the protocol, or interfere with the interpretation of the safety results;
* 11. Subjects with active, known, or suspected autoimmune disease. Subjects were eligible if they had type I diabetes, hypothyroidism requiring only hormone replacement therapy, skin conditions that did not require systemic treatment (such as vitiligo, psoriasis, or alopecia), or conditions that were not expected to recist in the absence of external stimuli;
* 12. All toxicities from previous anticancer treatment (except alopecia and fatigue) had to have returned to grade 1 (according to NCI CTCAE, version 4) or baseline before starting the study drug. Subjects were eligible if the toxicity of previous anticancer therapy was not expected to resolve and resulted in long-term sequelae, such as neuropathy after treatment with platinum-based agents
* 13. Subjects must have recovered from major surgery or severe trauma for at least 14 days before the first dose of study treatment;
* 14. Subjects who have received previous cellular immunotherapy such as cytokine-induced killer [CIK] therapy;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PS score 2 for locally advanced/advanced non-small cell lung cancer with negative driver genes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time | 2 year
  The time from the date of randomization to the date of first documented disease progression, assessed up to 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangdong, Guangzhou, China